CLINICAL TRIAL: NCT02008162
Title: Response to Bronchodilation With Tiotropium Plus Salbutamol Correlates With Radiologic Morphology of the Lung in COPD of the Emphysematous Phenotype
Brief Title: Bronchoreversibility and Radiologic Morphology of Emphysema
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Eugenio Pompeo, Associate Professor, University of Rome Tor Vergata
Other Study IDs: BREPTV-108.7
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Emphysema; COPD
Keywords: Emphysema, COPD, bronchoreversibility, ventilatory obstruction, lung volume reduction surgery, LVRS
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive | interventions — Bronchodilator Agents; Albuterol; Tiotropium Bromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bronchodilators: Patients with severe heterogeneous emphysema selected as potential candidtes for lung volume reduction surgery.
  Bronchodilators employed for the study include albuterol 200µg and tiotropium bromide 18 µg administered by puffs following a first spirometry and plethysmography performed after a washout period of 48h from all bronchodilators and subsequently repeated within 30 min after bronchodilators administration.
  Interventions: Drug: Bronchodilators

INTERVENTIONS:
Drug: Bronchodilators — Administration of both albuterol and tiotropium bromide after a 48h period of washout from all bronchodilators, followed by spirometry and plethysmography
  Other Names: Albuterol; Tiotropium bromide

SUMMARY:
To assess response to bronchodilation with tiotropium plus salbutamol in patients with severe emphysema and analyze relationships between bronchoreversibility response and semiquantitative computed-tomography based emphysema severity measures.

ELIGIBILITY:
Inclusion Criteria:

* Radiologic evidence of severe heterogeneous emphysema
* GOLD COPD class III-IV
* No other significant pulmonary comorbidity
* Quit smoking since at least 4 months

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe heterogeneous emphysema selected as potential candidtes for lung volume reduction surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-11; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
post-bronchodilator FEV1 change | 1 h
  Assessed by spirometry carried out before and after administration of bronchodilators
post-bronchodilator change in FVC | 1h
  Assessed by spirometry carried out before and after administration of bronchodilators

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Pompeo, MD, Principal Investigator — Tor Vergata University
Locations (1):
- Fondazione Policlinico Tor Vergata, Rome, Italy